CLINICAL TRIAL: NCT02014974
Title: INORMUS 5,000: Large Observational Study of Orthopedic Trauma Patients
Brief Title: InterNational ORthopaedic MUlticenter Study in Fracture Care
Acronym: INORMUS
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: McMaster Surgical Associates (Other)
Responsible Party: Principal Investigator, Mohit Bhandari, Professor of Surgery, Chair of Division of Orthopaedics, McMaster University
Other Study IDs: INORMUSINDIA
Record Dates: First submitted 2011-09-27; First posted 2013-12-19 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Bone Fractures
Keywords: Fractures; burden of fractures; orthopaedic fractures; orthopaedic injuries; orthopaedic trauma; fractures India; observational study; outcomes of fracture care; wait times India; epidemiology
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Public Hospitals: Patients presenting and treated in public trauma centers in India.
- Private Hospitals: Patients presenting and treated in private trauma centers in India.

SUMMARY:
Background: Worldwide injuries from trauma accidents represents a major population problem. The World Health Organization (WHO) has deemed this problem as one of the most important global priorities, calling 2011-2021 the Global Road Traffic Safety Decade. Despite this, there is little empirical data in low and middle-income countries quantifying the burden of fractures and the current practice of care.

Methods: The investigators conducted a multicenter, prospective observational study of patients sustaining fractures or dislocations who presented to an orthopaedic fracture unit at 14 hospitals in India. A representative sample of patients were recruited during an 8-week period starting on October 1, 2012. Patients were followed up to 30-days in hospital or until discharge to determine if they suffered any outcomes. Primary outcomes included total mortality, reoperation, and infection.

DETAILED DESCRIPTION:
INTRODUCTION

Global Epidemic of Trauma: Injuries from trauma accidents have been rapidly increasing in number worldwide and particularly so in developing countries. Approximately 5.8 million people die every year from traumatic injuries, accounting for 10% of the world's deaths. According to a recent report by the World Health Organization, trauma will be the third largest killer in the developing world by 2020. Moreover, for every death, several thousand individuals will suffer impairments, frequently with disabling consequences. Among the Southern Asian countries, India has the highest incidence of deaths due to physical injuries (117 deaths per 100,000 individuals). Physical injuries account for 10% of deaths, 20-25% of hospitalizations, and one third of disabilities. As this trend is growing, it is leading to an increase in the number of physical injury hospitalizations. Most developing nations, where trauma burden is escalating, have little empirical data on types of injuries, access to care, and management approaches. The investigators propose a prospective study in India (the second most populous country in the world) to examine fracture burden and provide the foundation for future collaboration and research. This study is fundamental to understanding the global burden of trauma and the design of future pragmatic randomized trials to improve function and quality of life around the world.

WHO Decade of Road Traffic Safety: This study directly aligns with the start of the Global Road Traffic Safety Decade 2011-2020 (World Health Organization), as well as our Department of Surgery's International Surgery Program. The Canadian Orthopaedic Association's 'call to action' to Canadian centers towards bridging gaps in knowledge and research in trauma in Low and Middle Income Countries further vindicates the rationale for INORMUS.

METHODS

Design Overview: Between October 2011 and March 2012, the investigators conducted a multicenter, prospective observational study of patients sustaining fractures and presenting to orthopaedic fracture units across 14 hospitals in India. 4,659 patients during an 8-week period were enrolled.

Patient characteristics, treatment, and outcome data were documented at initial consultation by a study coordinator at each hospital. Major complications, in hospital, and 30-day outcomes were evaluated.

Primary outcome

1. Logistic regression model involving 12 potential predictors of mortality;

   Secondary Analyses
2. Mixed-model involving the 12 predictors of mortality to evaluate potential hospital site effects;
3. Logistic regression model looking at timing of irrigation and debridement and open fractures and deep infection rates;
4. Descriptive analyses looking at types of treatments of tibia and femur fractures across socioeconomic groups in India;
5. Descriptive analyses looking at combinations of injuries in patients involved in road traffic accidents.

Sample Size: The study enrolled 4,822 patients, and 4,612 (95.6%) of these patients completed follow-up. To include 12 predictors in the model with an estimated mortality rate among orthopedic trauma patients of 1.5%, 8000 patients are required to properly power our analysis. Based on a 20% drop out rate, 10,000 patients will be recruited in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Over 17 years old;
2. Diagnosis of orthopaedic fracture or dislocation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We have planned a multicenter, prospective observational study of patients sustaining fractures and presenting to orthopaedic fracture units across hospitals in India. All patients with an orthopaedic injury presenting participating hospitals during an 8-week period will be approached for study enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 4822 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
30-day Mortality | 30 days post injury
  Logistic regression including 12 a priori predictors of mortality.

SECONDARY OUTCOMES:
Deep Infection | 30 days post-injury
  Logistic regression including 8 a priori predictors of deep infection in open fracture patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD, PhD, Principal Investigator — McMaster; Parag Sancheti, MD, Study Director — Sancheti Institute for Orthopaedics
Locations (1):
- Sancheti Institute of Orthopaedics, Pune, Maharashtra, India

REFERENCES:
- [Background] Rodgers A, Ezzati M, Vander Hoorn S, Lopez AD, Lin RB, Murray CJ; Comparative Risk Assessment Collaborating Group. Distribution of major health risks: findings from the Global Burden of Disease study. PLoS Med. 2004 Oct;1(1):e27. doi: 10.1371/journal.pmed.0010027. Epub 2004 Oct 19. PMID 15526049
- [Background] Stone DH, Gofin R. The 8th World Conference on injury prevention and safety promotion. Inj Prev. 2007 Feb;13(1):70. doi: 10.1136/ip.2006.014001. No abstract available. PMID 17296697
- [Background] Joshipura MK. Trauma care in India: current scenario. World J Surg. 2008 Aug;32(8):1613-7. doi: 10.1007/s00268-008-9634-5. PMID 18553048
- [Background] Joshipura M. Guidelines for essential trauma care: progress in India. World J Surg. 2006 Jun;30(6):930-3. doi: 10.1007/s00268-005-0765-7. PMID 16736317
- [Background] Joshipura MK, Shah HS, Patel PR, Divatia PA, Desai PM. Trauma care systems in India. Injury. 2003 Sep;34(9):686-92. doi: 10.1016/s0020-1383(03)00163-3. PMID 12951294
- [Background] Mock C, Cherian MN. The global burden of musculoskeletal injuries: challenges and solutions. Clin Orthop Relat Res. 2008 Oct;466(10):2306-16. doi: 10.1007/s11999-008-0416-z. Epub 2008 Aug 5. PMID 18679760
- [Background] Ma ZS, Zhang HJ, Lei W, Xiong LZ. Musculoskeletal trauma services in China. Clin Orthop Relat Res. 2008 Oct;466(10):2329-36. doi: 10.1007/s11999-008-0382-5. Epub 2008 Jul 16. PMID 18629598
- See also: United Nations Global Road Traffic Safety Collaboration — http://www.who.int/roadsafety/en/
- See also: Canadian Orthopaedic Association: Call for Action Group — http://www.coa-aco.org/
- See also: WHO's Make Roads Safe Campaign — http://www.makeroadssafe.org/Pages/home.aspx
- See also: McMaster University International Surgery Desk — http://www.makeroadssafe.org/Pages/home.aspx